CLINICAL TRIAL: NCT06599866
Title: Turkish Validity and Reliability of the Core Lower Urinary Tract Symptoms Questionnaire in Patients With Multiple Sclerosis
Brief Title: Turkish Validity and Reliability of the Core Lower Urinary Tract Symptoms Questionnaire in Individuals With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/04-13
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Lower Urinary Track Symptoms; Multiple Sclerosis
Keywords: lower urinary tract symptoms; multiple sclerosis; reliability; validity
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Sclerosis Group: Individuals between the ages of 18-65 who have been diagnosed with multiple sclerosis by a specialist physician.

SUMMARY:
The aim of this study is to study the validity and reliability of Core Lower Urinary Tract Symptoms Score in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis is an autoimmune disease that can affect any part of the central nervous system. Multiple sclerosis, whose prevalence is increasing every year in the world, brings with it many symptoms. Lower urinary tract symptoms develop secondary to demyelinating lesions in the spinal cord and pontine micturition center in the disease pathophysiology commonly seen in Multiple sclerosis and other symptoms seen in Multiple sclerosis (inactivity, fear of movement, etc.). Due to the multifocal and widespread involvement of the CNS, Lower urinary tract symptoms in Multiple sclerosis patients are variable and their severity varies among Multiple sclerosis patients. Lower urinary tract symptoms are divided into 3 groups as storage, voiding and post-voiding symptoms. The rate of urinary complications in Multiple sclerosis patients is significantly higher compared to the general population. Although it is a common symptom in multiple sclerosis , the evaluation of Lower urinary tract symptoms in individuals with Multiple sclerosis is quite limited in the literature. Evaluation of Lower urinary tract symptoms seen in Multiple sclerosis with appropriate assessment tools is important to obtain comprehensive information about the progression of the disease. There are many questionnaires used in the evaluation of Lower urinary tract symptoms. While the International Prostate Symptom Score and the Danish Prostate Symptom Score, which are frequently used for benign prostatic hyperplasia, are used; Overactive Bladder Questionnaire-V8 was developed to evaluate overactive bladder symptoms. However, these questionnaires are also frequently used in the evaluation of Lower urinary tract symptoms. Since the purpose of developing the questionnaires is for different diseases, they are not comprehensive enough for Lower urinary tract symptoms. The Core Lower Urinary Tract Symptoms Score is a questionnaire developed to comprehensively evaluate lower urinary tract symptoms. Although the Core Lower Urinary Tract Symptoms Score Turkish validity and reliability study was conducted by Erbay et al. in 2022, its validity and reliability in Multiple sclerosis patients has not been performed.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years old
* Being diagnosed with multiple sclerosis by a specialist
* Being willing to participate in the study
* Being literate

Exclusion Criteria:

* Not volunteering to participate in the study
* Having a neurological disorder that prevents speech

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being diagnosed with multiple sclerosis by a specialist physician between the ages of 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Core Lower Urinary Tract Symptoms Score | 10 minuttes
  The questionnaire was developed by Homma et al. in 2008 to assess lower urinary tract symptoms. The Turkish validity and reliability study of the questionnaire was conducted by Erbay et al. in 2022. The first 5 questions in the 13-question questionnaire are about storage problems, the next 3 questions are about urination problems, and the next 2 questions are about lower urinary tract pain. The first 10 questions are scored on a Likert-type scale from 0 to 3. The Core Lower Urinary Tract also includes a question asking participants to list three core symptoms (question 11) and a question about the primary core symptom (question 12). It also includes a question about quality of life (question 13). The last question is about the patients' satisfaction with their current urinary status, scored from 0 to 6.

SECONDARY OUTCOMES:
Overactive Bladder Questionnaire-V8 | 5 minutes
  Overactive Bladder Questionnaire was first developed in English by Coyne and colleagues in 2002. In later studies, Overactive Bladder Questionnaire short form and shorter forms such as Overactive Bladder Questionnaire-V8 were developed. Overactive Bladder Questionnaire-V8 consists of the first 8 questions of Overactive Bladder Questionnaire and was recommended as an Overactive Bladder Questionnaire screening and awareness test. The validity and reliability of the questionnaire in Turkish was conducted by Tarcan et al. in 2012. Today, it is frequently used to evaluate lower urinary tract symptoms. The Overactive Bladder Questionnaire-V8 uses a Likert-type scale of 0-5 to determine the severity of individuals' complaints: None (0); a little (1); a little (2); a lot (3); a lot (4); a lot (5). The total score is between 0 and 40. If the total score obtained from the questionnaire is more than 8, individuals are considered to have possible lower urinary tract symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiloatar H, Delibay AA, Demir CO, Ceylan D, Uysal N. Reliability and validity of the Turkish version of the core lower urinary tract symptom score in multiple sclerosis. Acta Neurol Belg. 2025 Jun;125(3):811-817. doi: 10.1007/s13760-025-02769-0. Epub 2025 Mar 26. PMID 40133731